CLINICAL TRIAL: NCT05507164
Title: Non-randomized Pilot Study to Characterize Temporo-masseteric Nerve Block (TMNB) in
Brief Title: Characterization of the Temporo-masseteric Nerve Block (TMNB) in Healthy Subjects
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Gayathri Subramanian, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro2022000182
Record Dates: First submitted 2022-08-11; First posted 2022-08-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Occlusion
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Temporo-masseteric Nerve Block Administration (Other): Non-randomized administration of the TMNB injection (unilateral) followed by bite force distribution and surface EMG assessment of the temporalis and masseter muscles on the side of the injection
  Interventions: Drug: Temporomasseteric Nerve Block

INTERVENTIONS:
Drug: Temporomasseteric Nerve Block — The TMNB injection is a local anesthetic injection technique that targets the anterior deep temporal and masseteric branches of the mandibular division of the Trigeminal Nerve. The surface landmark for the twin block injection site is located by palpating for the depression created by the greater wing of the sphenoid bone at the superior border of the zygomatic process and approximately 1 cm posterior to the posterior border of the frontal process of the zygomatic bone. This site is first disinfected with alcohol wipes prior to inserting a 27- or 25-gauge long dental needle (32 mm). Angled 35-45° away from the calvarium (skull) and perpendicular to the zygomatic arch (along the coronal plane), the needle is advanced to its length before injecting 1.8 mL of 2% lidocaine with 1:100,000 epinephrine.
  Other Names: Twin Block

SUMMARY:
The proposed pilot study is aimed at preliminary characterization of the TMNB injection in 20 healthy volunteers. Assessment of bite-force distribution and surface electromyographic activity of the temporalis and the masseter muscles, at rest and clench, before and after unilateral TMNB injection, will be the primary outcome measures. Post-injection assessments will be performed at 30 minutes, 2 hours, and 2 weeks after the injection. Participants will be surveyed regarding their experience receiving the TMNB injection (secondary outcomes).

DETAILED DESCRIPTION:
1.1 Purpose/Specific Aims The Temporo-masseteric Nerve Block (TMNB) is a local anesthetic injection targeting the deep temporal and masseteric branches of the mandibular division of the Trigeminal Nerve, that supply the temporalis and masseter muscles. Emerging evidence supports the TMNB's therapeutic potential in alleviating both acute and chronic myogenous pain of temporalis or masseteric origin. The TMNB injection is safe and well tolerated by patients.

The nerves targeted by the TMNB are mixed nerves and supply both sensory and motor innervation to the muscles. In addition, pain relief from the TMNB injection is sustained beyond the duration of the local anesthetic's duration of action. It is important to characterize the TMNB block, particularly its effects on the target muscles to understand the mechanism for its sustained pain relief.

The temporalis and the masseter muscles mediate jaw closure and clenching actions. The proposed pilot study is aimed at preliminary characterization of the TMNB injection in 20 healthy volunteers. Assessment of bite-force distribution and surface electromyographic activity of the temporalis and the masseter muscles, at rest and clench, before and after unilateral TMNB injection, will be the primary outcome measures. Post-injection assessments will be performed at 30 minutes, 2 hours, and 2 weeks after the injection. Participants will be surveyed regarding their experience receiving the TMNB injection (secondary outcomes).

A. Objectives The proposed pilot study is aimed at preliminary characterization of the TMNB injection in 20 healthy volunteers. Assessment of bite-force distribution and surface electromyographic activity of the temporalis and the masseter muscles, at rest and clench, before and after unilateral TMNB injection, will be the primary outcome measures. Post-injection assessments will be performed at 30 minutes, 2 hours, and 2 weeks after the injection. Participants will be surveyed regarding their experience receiving the TMNB injection (secondary outcomes).

B. Hypotheses / Research Question(s) (Alternate hypotheses)

1. The TMNB injection alters bite force distribution
2. The TMNB injection alters the surface electromyographic activity of the temporalis and masseter muscles on the side of the injection

1.2 Research Significance The TMNB injection is a local anesthetic injection technique that targets the anterior deep temporal and masseteric branches of the mandibular division of the Trigeminal Nerve. It has been in clinical use for over seven years. It has value as a diagnostic tool in helping differentiate between a toothache and jaw muscle pain when it is difficult for the patient and the clinician to otherwise differentiate between the two. In addition, it also has the ability to ease chronic jaw muscle pain that impacts the masseter and temporalis muscles. However, the mechanism of its sustained pain relief is not known. Given that the local anesthetic action usually lasts for over an hour, it is important to decipher how the TMNB brings about sustained pain relief for longer periods of time. In fact, the pain relief achieved by the TMNB injection in chronic myogenous Temporomandibular disorder involving the masseter and temporalis muscles is comparable to trigger point injections, a standard management modality that requires specialty training and hence is not readily accessible to all patients. The investigators speculate that the nerves to the masseter and temporalis muscles being mixed nerves (i.e., carrying both sensory and motor nerve supply), administration of the TMNB injection could ease muscle tone and activity, relieving chronic pain. Interruption of the pain-contraction-pain cycle may help relieve chronic pain. In order to verify this speculation, the investigators propose the use of TMNB in healthy subjects followed by assessment of jaw muscle function, as measured by bite force distribution and surface electromyographic assessment of the masseter and temporalis muscles. Elucidating the mechanism of TMNB's action has important implications on understanding its therapeutic potential in mTMD as well as elucidating the mechanisms of chronic myogenous TMD itself.

1.3 Research Design and Methods This study is a non-randomized prospective pilot study with twenty study subjects. Assessment of bite-force distribution and surface electromyographic activity of the temporalis and the masseter muscles, at rest and clench, before and after unilateral TMNB injection, will be the primary outcome measures. Post-injection assessments will be performed at 30 minutes, 2 hours, and 2 weeks after the injection, to capture the impact of onset, known duration of action of the local anesthetic used for the study (standard dental local anesthetic, 2% lidocaine with 1:100,000 epinephrine) after a period of 2 weeks.5 Participants will be surveyed regarding their experience receiving the TMNB injection (secondary outcomes).

A. Research Procedures The study will be conducted at the Clinical Research Center at Rutgers School of Dental Medicine. Healthy subjects with no history of TMDs will be recruited (see Eligibility criteria, Figure 1a and b).6 10 male and 10 female subjects will be recruited as per criteria outlined elsewhere.

Subject eligibility and initial evaluation will be conducted by PI SA, a Board-certified Oro-facial Pain Specialist. Informed consent will be obtained from all study participants and all participants can withdraw study consent at any time during the study. The TMNB injection will be delivered using the published technique. The needle position will be verified using a Nerve conduction study (a standard technique for verification of motor nerve blocks). The subsequent assessments including occlusal analysis (OA) and surface electromyography (sEMG) will be administered by either PI GS, PI SA or Co-I SYPQ, using T-scan/BioEMG (Tekscan, Inc., Boston, MA and BioRESEARCH, Inc., Brown Deer, WI). The side of TMNB administration will randomly assigned as left or right side.

Participants will be surveyed regarding their experience receiving the TMNB injection (secondary outcomes). The questionnaire will be offered to the subjects on the day of their injection and again at the two-week post-TMNB injection.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years of age
* All ethnicity
* Male and female sex
* Fluent in written/spoken English
* Never been diagnosed with TMD
* No significant history of orofacial pain
* <5 headaches/month in the 3 months before enrollment
* No reported use of a nightguard or occlusal splint 'No' to all questions on self-administered questionnaire for TMD screening:
* Pain in jaw or temple on either side of the face in the last 30 days
* Stiffness or pain in jaw upon awakening in the last 30 days
* Any pain increase/reduction in the jaw/temple region during the last 30 days with

  * Chewing hard or tough food
  * Opening mouth or moving jaw forward or to the side
  * Hold teeth together/clenching/grinding/chewing gum
  * Using the jaw during activities such as talking, kissing or yawning

Exclusion Criteria:

* Traumatic injury/ surgery on face or jaw < 6 months
* current orthodontic treatment
* pregnant or nursing,
* kidney failure or renal dialysis,
* heart disease or heart failure,
* uncontrolled chronic respiratory disease/ hypertension/ diabetes
* history of
* seizures
* hyperthyroidism
* drug or alcohol abuse
* psychiatric disorder/conditions requiring hospitalization
* chemotherapy/radiation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 10 males and 10 female subjects will be enrolled in the study
Enrollment: 20 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Bite force distribution | Baseline, 30 min, 2 hours and 2 weeks
  Left vs Right distribution of bite force upon clenching will be assessed as an average of 3 consequent measurements.
Change in Surface EMG | Baseline, 30 min, 2 hours and 2 weeks
  Surface EMG will be utilized to measure surface electrical activity over the temporalis and masseter muscles at rest and clenching
Survey | At 2 weeks post injection
  All subjects will be surveyed for their experience as part of their participation in the study

CONTACTS AND LOCATIONS:
Overall Officials: Gayathri D Subramanian, DMD, Principal Investigator — Rutgers School of Dental Medicine
Locations (1):
- Rutgers School of Dental Medicine, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
After study completion, deidentified data can be shared.
Supporting Information: Study Protocol, CSR
Time Frame: Within 4 weeks of approved request after study completion, at time of publication
Access Criteria: By individual request

REFERENCES:
- [Background] Quek S, Young A, Subramanian G. The twin block: a simple technique to block both the masseteric and the anterior deep temporal nerves with one anesthetic injection. Oral Surg Oral Med Oral Pathol Oral Radiol. 2014 Sep;118(3):e65-7. doi: 10.1016/j.oooo.2014.01.227. Epub 2014 Feb 6. PMID 24703404
- [Background] Ananthan S, Kanti V, Zagury JG, Quek SYP, Benoliel R. The effect of the twin block compared with trigger point injections in patients with masticatory myofascial pain: a pilot study. Oral Surg Oral Med Oral Pathol Oral Radiol. 2020 Mar;129(3):222-228. doi: 10.1016/j.oooo.2019.09.014. Epub 2019 Oct 13. PMID 32009005
- [Background] Quek SYP, Kalladka M, Kanti V, Subramanian G. A new adjunctive tool to aid in the diagnosis of myogenous temporomandibular disorder pain originating from the masseter and temporalis muscles: Twin-block technique. J Indian Prosthodont Soc. 2018 Apr-Jun;18(2):181-185. doi: 10.4103/jips.jips_293_17. PMID 29692573
- [Background] Kanti V, Ananthan S, Subramanian G, Quek SYP. Efficacy of the twin block, a peripheral nerve block for the management of chronic masticatory myofascial pain: A case series. Quintessence Int. 2017 Oct 6:725-729. doi: 10.3290/j.qi.a39094. Online ahead of print. PMID 28990015
- [Background] Schiffman E, Ohrbach R. Executive summary of the Diagnostic Criteria for Temporomandibular Disorders for clinical and research applications. J Am Dent Assoc. 2016 Jun;147(6):438-45. doi: 10.1016/j.adaj.2016.01.007. Epub 2016 Feb 26. PMID 26922248
- [Background] Quek SYP, Gomes-Zagury J, Subramanian G. Twin Block in Myogenous Orofacial Pain: Applied Anatomy, Technique Update, and Safety. Anesth Prog. 2020 Jun 1;67(2):103-106. doi: 10.2344/anpr-67-01-03. PMID 32633773